CLINICAL TRIAL: NCT00818194
Title: A Comparison of Effects of Short-term Low Dose Exposure of Advagraf® and Neoral® Microemulsion Cyclosporine A on Renal Perfusion and Function in Healthy Volunteers
Brief Title: Comparison of Extended Release Tacrolimus (Advagraf) and Cyclosporine A Microemulsion on Renal Function in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FKC-012; Health Canada Control # 119562
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Tacrolimus; cyclosporine A; renal plasma flow; glomerular filtration rate; human; pharmacodynamics; pharmacokinetics; Pharmacodynamics of tacrolimus
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. tacrolimus first (Experimental): Subjects receive extended release tacrolimus in first dosing interval then cross over to cyclosporine A for second dosing interval
  Interventions: Drug: extended release tacrolimus; Drug: cyclosporine A microemulsion
- B. cyclosporine first (Experimental): Subjects receive cyclosporine A in first dosing interval then cross over to extended release tacrolimus for second dosing interval
  Interventions: Drug: extended release tacrolimus; Drug: cyclosporine A microemulsion

INTERVENTIONS:
Drug: extended release tacrolimus — oral
  Other Names: Advagraf®; FK506E; MR4
Drug: cyclosporine A microemulsion — oral
  Other Names: Neoral®

SUMMARY:
The purpose of this study is to compare the effects of steady state tacrolimus vs. cyclosporine on renal pharmacodynamics in healthy volunteers.

DETAILED DESCRIPTION:
This study seeks to evaluate the renal physiological responses of short-term maintenance level doses of CNIs in healthy volunteers to determine if daily perturbations in renal physiology exist, and if confirmed, whether they differ between CNIs and thus may contribute by different mechanisms to the progression of CAN.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* healthy with no history or current clinical findings of infection or disease of the following nature: cerebrovascular, neurologic, cardiovascular, endocrine, pulmonary, immunologic, metabolic, hematologic, diabetes mellitus, glucose intolerance, gout
* non-smoker and willing to abstain from alcohol consumption during the study
* agrees to use appropriate contraception during the study period until 3 months after the final study exam.

Exclusion Criteria:

* history of significant alcohol abuse or drug abuse within 1 year prior to the screening visit
* regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week)
* use of soft drugs (marijuana) within 3 months prior to the screening visit or hard drugs (cocaine, PCP, crack) within 1 year prior to the screening visit Hepatitis B or C, HIV, history of cancer (excluding excised squamous or basal cell carcinoma)
* positive tuberculin skin test or prior TB infection
* known history of serious head injuries, seizures or any eating disorder
* received an investigational drug within 30 days prior to the first study drug administration
* known hypersensitivity/allergy to tacrolimus, cyclosporine, iothalamate iodine, para-aminohippuric acid, antibiotics or antifungals
* Body mass index (BMI) <19 or >27
* clinically significant history of psychiatric disease or a significant disability that prevents understanding or adherence to protocol
* renal dysfunction, serum creatinine or urine microalbumin above the normal age and gender-adjusted reference range of the local lab
* clinically significant abnormal liver function test indicative of impaired hepatic function
* received medications/herbal preparations that may affect the metabolism of tacrolimus or cyclosporine A within 1 month of the first study drug administration
* received any other prescription medication within 14 days prior to the first study drug administration or any over-the-counter product within 7 days prior to the first study drug administration, except for topical products without systemic absorption
* current GI condition known to affect GI motility and/or absorption
* donation of plasma (500 mL) within 7 days prior to the first study drug administration or donation/ loss of whole blood as follows: 50 mL to 499 mL within 30 days or more than 499 mL within 56 days prior to the first study drug administration
* clinically significant surgery within 4 weeks prior to the first study drug administration
* administration of steroids by injection within 12 weeks prior to the first study drug administration
* administration of any live vaccine within 7 days prior to the first study drug administration
* travel in areas where TB is endemic within 8 weeks prior to the TB skin test performed at the screening visit
* hemoglobin <140 g/L

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Effective Renal Plasma Flow response | Baseline and Day 10 of each dosing interval

SECONDARY OUTCOMES:
Comparison of Glomerular Filtration Rate response | Baseline and Day 10 of each dosing interval
Comparison of blood pressure response | Baseline and Day 10 of each dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (1):
- Montreal, Quebec, Canada